CLINICAL TRIAL: NCT07391839
Title: A Multicenter, Open-label, Single-Arm Phase I/II Clinical Study to Evaluate the Safety and Efficacy of a Single Dose of MDN-001 Injection in Patients With Unresectable Primary Hepatocellular Carcinoma (HCC).
Brief Title: MDN-001 Injection for the Treatment of Unresectable Primary Hepatocellular Carcinoma.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Mednovo Yi Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDN-001
Record Dates: First submitted 2025-12-17; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-04

CONDITIONS: Hepatoma; Unresectable Hepatocellular Carcinoma (HCC)
Keywords: unresectable hepatocellular carcinoma; HCC; Yttrium-90 Microsphere
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDN-001 Injection(Yttrium-90 Microsphere Injection) (Experimental)
  Interventions: Drug: MDN-001 Injection(Yttrium-90 Microsphere Injection)

INTERVENTIONS:
Drug: MDN-001 Injection(Yttrium-90 Microsphere Injection) — Yttrium-90 Microsphere Injection

SUMMARY:
The main purpose of the study is to evaluate the safety and efficacy of MDN-001 injection(Yttrium-90 Microsphere Injection)in the treatment of unresectable hepatocellular carcinoma. Other purposes of this study include assessment of the effect of treatment on overall survival, the length of time it takes for the disease to worsen, if and how the treatment affects the patient's quality of life, and if and how the cancer responds to the treatment.

DETAILED DESCRIPTION:
A multicenter, open and single-arm phase I clinical study to evaluate the safety and efficacy of MDN-001 injection(Yttrium-90 Microsphere Injection) in the treatment of unresectable hepatocellular carcinoma. The study aims to recruit 40 patients over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to join this study and sign the informed consent form.
* Age: 18~80 years old (inclusive), regardless of gender.
* Clinically diagnosed hepatocellular carcinoma or pathologically diagnosed hepatocellular carcinoma.
* ECOG performance status of 1 or less
* Child-Pugh score A or better B (≤7).
* Patients who are assessed by researchers as currently unacceptable for surgical resection or ablation, or who refuse to undergo surgical resection or ablation.
* According to mRECIST standard, in contrast-enhanced MRI or CT images, there must be at least one measurable liver target lesion with the longest diameter ≥1 cm. If there are multiple target lesions, the researcher will choose them.
* According to the researcher's evaluation, the expected survival time is ≥3 months.
* There is no extrahepatic metastasis, and there are no other malignant tumors besides liver cancer.
* The main organs function normally and meet the following requirements: blood routine: no blood transfusion or colony stimulating factor (G-CSF) treatment within 14 days before signing the informed consent form, and hemoglobin ≥ 80g/L; Platelet count > 50× 109/L; Neutrophil count (ANC) ≥ 1.5× 109/L. Liver function: serum total bilirubin (TBIL)≤2 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤5.0 times ULN；; Alkaline phosphatase (ALP)≤2.5 times ULN；; Albumin > 30 g/L. Renal function: creatinine (Cr)≤1.5 times ULN；; Creatinine clearance rate ≥50 mL/min (calculated according to Cockcroft-Gault formula). Coagulation function: INR, PT and APTT)≤1.5 times ULN. If the subjects take warfarin or heparin for anticoagulant therapy, it is necessary to ensure that they meet the requirements of the protocol when they stop taking the drug or not. Cardiovascular function: echocardiography: LVEF (left ventricular ejection fraction) ≥50%.
* According to the standard of CTCAE5.0, all the adverse events of previous systemic anti-tumor therapy were restored to baseline or ≤1 grade [except: the neuropathy induced by previous anti-tumor therapy was stable (≤2 grade); Hair loss, fatigue, etc., which are judged by the researchers based on the actual clinical situation, cannot be restored to ≤1 level and will be in a stable state for a long time; Stable hypothyroidism after hormone replacement therapy].
* Women and men of childbearing age must agree to take strict and effective contraceptive measures after signing informed consent, during the study period and within 6 months after the end of the experiment; Men are forbidden to donate sperm during this period, and the pregnancy test results of female subjects of childbearing age during the screening period and within 24 hours before administration must be negative.

Exclusion Criteria:

Participants who meet any of the following criteria are not allowed to participate in this study:

* Severe liver dysfunction: including severe jaundice, hepatic encephalopathy, refractory ascites or hepatorenal syndrome.
* Patients who are suitable for surgical resection or ablation after evaluation by researchers: 1) patients who are suitable for surgical resection include but are not limited to the following situations: a) patients with good liver reserve function in CNLC Ia~IIa stage; B) If the tumor is confined to the same hepatic segment or ipsilateral hemihepatis, after MDT discussion, the patients with CNLC IIb stage who may get better effect by surgical resection than other treatments; 2) Suitable for ablation treatment includes but is not limited to the following situations: A)CNLC Ia patients; B) patients with CNLC Ib stage and Child-Pugh score of liver function grade A or better grade B (≤7).
* The liver area has received external radiotherapy before.
* Severe pulmonary insufficiency (FEV1/FVC&1t; 50% or FEV1&1t: 50% expected value or maximum ventilation per minute < 50 L/min), patients with obvious chronic obstructive pulmonary disease or interstitial pneumonia.
* Arterial perfusion imaging of technetium [99mTc] polymerized albumin (99mTc-MAA) showed that the percentage of hepatopulmonary shunt was more than 20%, or the absorbed dose of single lung radiation was more than 30 Gy, or the accumulated absorbed dose of lung radiation was more than 50 Gy.
* Hepatic arteriography and 99mTc-MAA hepatic artery perfusion imaging showed gastrointestinal shunts, which may not be corrected by vascular interventional techniques.
* Can't intubate hepatic artery, such as vascular malformation, allergic to contrast agent, allergic to anesthetic, etc.
* There is a tumor thrombus in the main portal vein.
* The last anti-tumor treatment (surgery, chemotherapy, immunotherapy, targeted therapy, etc.) is less than 4 weeks before the administration of the experimental drug.
* Participation in other clinical studies within 4 weeks before the first administration of the study drug.
* It is expected that any other forms of anti-tumor therapy will be needed during the study.
* Those who have been vaccinated with live attenuated vaccine within 28 days before the administration of the first study drug or plan to be vaccinated within 60 days after the treatment of the study drug.
* People with previous history of epilepsy.
* Patients who have undergone major organ surgery (excluding puncture biopsy) or had significant trauma within 4 weeks before the first use of the study drug, or need to undergo elective surgery during the trial.
* Patients who have undergone bone marrow transplantation or solid organ transplantation in the past.
* Untreated or being treated tuberculosis patients, including but not limited to tuberculosis; Those who have been treated with standardized anti-tuberculosis treatment and confirmed to have been cured by researchers can be included.
* Patients with active infection of grade ≥2 who need systemic treatment of antibiotics within 2 weeks before the administration of the study drug.
* Patients who have been diagnosed with immunodeficiency disease and/or who have tested positive for human immunodeficiency virus (HIV) at the time of screening.
* Patients with clinically significant cardiovascular and cerebrovascular diseases within 6 months before the first administration of the study drug, including but not limited to: acute myocardial infarction; Severe/unstable angina pectoris; History of arterial thromboembolism, including but not limited to cerebrovascular accidents; Congestive heart failure [new york Heart Association (NYHA) > Grade II; Any clinically significant resting ECG rhythm, abnormal conduction or morphology, complete left bundle branch block, degree III cardiac block, degree II cardiac block, and PR interval > 250 ms；; The average corrected QT interval (QTCF) obtained by three ECG examinations is > 450 msec (C male) or > 470 msec (female) (only when the first ECG prompts QTCF to be > 450 msec (male) or > 470 msec (female), it is necessary to retest and take the average corrected value for three times (corrected according to Fridericia formula); Hypertension beyond the control of antihypertensive drugs (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg). Other cardiovascular and cerebrovascular diseases that researchers think are not suitable for selection.
* Have a history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonia requiring steroid treatment, or any evidence of clinically active ILD.
* Patients with mental illness that is known to interfere with trial compliance or still need drug control.
* Pregnant or lactating female patients.
* Any patient with severe, acute or chronic medical or mental illness or laboratory abnormality who may increase the risk of participating in the study or using the study drugs or may interfere with the interpretation of the study results and who the researcher thinks will not be suitable for participating in the study.
* According to the investigator's judgment, any other circumstances that prevent the patient from participating in the clinical trial (for safety reasons) or hinder the compliance of the clinical trial procedure (for example, difficulty in venous blood collection).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Type, frequency, and severity of adverse events (AEs), serious adverse events (SAEs), treatment-emergent adverse events (TEAEs), and treatment-related adverse events (TRAEs) | 12 months
  Record the types, frequencies and severity of AEs, SAEs, TEAEs and TRAEs, and grade them according to CTCAE v5.0.
Objective remission rate（IRC） | 6 months
  The objective remission rate of liver target lesions evaluated by independent review committee (IRC) 6 months after administration of MDN-001 injection.
Blood biochemistry (including ALT, AST, ALP, Cr and CCr) | 12 months
CBC (including WBC, RBC and Hb) | 12 months
Urinalysis (including BLD, BIL and PRO) | 12 months
Coagulation function (including PT andAPTT) | 12 months
Cardiac enzyme panel (including CK, CK-MB and cTn) | 12 months
Stool examination and OB | 12 months
12-lead ECG | 12 months
  OT interval (milliseconds), Rate (times per minute)
Vital signs | 12 months
  Body temperature (℃), Pulse/Heart rate (beats per minute, bpm)
Weight and Height | 12 months
  Weight in kilograms and height in meters

SECONDARY OUTCOMES:
Objective remission rate | 12 months
  (According to mRECIST and RECIST v1. 1 standards)Objective remission rate of liver target lesions assessed by researchers.
Time to disease progression | 12 months
  (According to mRECIST and RECIST v1. 1 standards)The time from liver target lesion to disease progression evaluated by researchers and IRC
Tumor Response Rate | 12 months
  (According to mRECIST and RECIST v1. 1 standards)The duration of remission (DOR), disease control rate (DCR) and complete remission rate (CRR) are evaluated by the researchers and IRC.
Progressively free survival | 12 months
Overall survival | 12 months
Changes of tumor marker alpha-fetoprotein before and after administration | 12 months
Actual distribution of yttrium-90 | 24 hours
  Actual distribution of yttrium -90 in human body within 24 hours after administration.
Radioactivity of Yttrium-90 in blood, urine and feces of Participants | 14 days
  Radioactivity of Yttrium -90 in blood, urine and feces of subjects after administration.
Absorbed dose and effective dose of internal irradiation after administration | 24 hours
  Absorbed dose and effective dose of internal irradiation after administration: The tumor/normal liver uptake ratio (T/N ratio) and liver shunt fraction (LSF) were calculated according to SPECT/CT or PET/CT data.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Zhongda Hospital, Nanjing, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Henan Cancer Hospital, Henan, Zhengzhou
  - Zhongshan hospital, Shanghai